CLINICAL TRIAL: NCT06788652
Title: Non-interventional Cohort Study of Patients Treated With Lisocabtagene Maraleucel (Liso-cel) for Relapsed/Refractory Mantle Cell Lymphoma in the Post-Marketing Setting
Brief Title: A Study of Patients With Relapsed/Refractory Mantle Cell Lymphoma Treated With Lisocabtagene Maraleucel in the Post-Marketing Setting
Status: Recruiting | Type: Observational
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CA082-1093
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants treated with lisocabtagene maraleucel
  Interventions: Biological: Lisocabtagene maraleucel

INTERVENTIONS:
Biological: Lisocabtagene maraleucel — According to US Prescribing Information

SUMMARY:
The purpose of this study is to understand the long-term safety and effectiveness of lisocabtagene maraleucel (liso-cel) for the treatment of Mantle Cell Lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

• Participants must have been treated in the postmarketing setting with at least 1 infusion of lisocabtagene maraleucel (Liso-cel) used for the treatment of Mantle Cell Lymphoma (MCL) according to the FDA-approved indication and dose range (ie, per the US Prescribing Information) and with a product meeting the specifications for commercial release approved in the USA

Exclusion Criteria:

* Participants known to be participating in investigational studies at the time of liso-cel infusion.
* Participants treated with non-conforming CAR T-cell product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults diagnosed with Relapsed/Refractory Mantle Cell Lymphoma (MCL) who are registered within the Center for International Blood and Marrow Transplant Research (CIBMTR) registry and have been treated with lisocabtagene maraleucel.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2044-09-30 (Estimated); Study Completion 2044-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 15 years

SECONDARY OUTCOMES:
Complete remission rate (CRR) | Up to 15 years
Overall response rate (ORR) | Up to 15 years
Progression-free survival (PFS) | Up to 15 years
Overall survival (OS) | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Center for International Blood and Marrow Transplant Research (CIBMTR), Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts